CLINICAL TRIAL: NCT05473832
Title: Evaluation of the Anti-aging Efficacy of Four Cosmetic Products
Brief Title: Evaluation of the Anti-aging Efficacy of Four Skin Health Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22.0229-39
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Anti-Aging; Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental)
  Interventions: Other: Day Cream cosmetic product compared to untreated side
- Group 2 (Experimental)
  Interventions: Other: Night cream cosmetic product compared to untreated side
- Group 3 (Experimental)
  Interventions: Other: Eye cream cosmetic product compared to untreated side
- Group 4 (Experimental)
  Interventions: Other: Serum cosmetic product compared to untreated side

INTERVENTIONS:
Other: Day Cream cosmetic product compared to untreated side — Applied once daily in the morning
  Arms: Group 1
Other: Night cream cosmetic product compared to untreated side — Applied once daily in the evening
  Arms: Group 2
Other: Eye cream cosmetic product compared to untreated side — Applied twice daily in the morning and in the evening around the eye area
  Arms: Group 3
Other: Serum cosmetic product compared to untreated side — Applied twice daily in the morning and in the evening
  Arms: Group 4

SUMMARY:
The purpose of this study is to assess the anti-wrinkle and anti-aging efficacy of four different cosmetic products compared to an untreated control (split-face study design)

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent to participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits
* Female and male
* From 40 to 65 years of age
* BMI < 30 kg/m2
* Healthy skin in the test areas
* Uniform skin color and no erythema or dark pigmentation in the test area
* Visible wrinkle in the face (grade 3 to 6 according to proderm scale) see Appendix 2
* Ethnicity: at least one Black, Asian and Hispanic subject per study group

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Active skin disease at the test area
* Documented allergies to face/eye care products
* Diabetes mellitus
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension (if not adjusted with medication), cardiovascular diseases
* Epilepsy
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, freckles, etc. at the test area that could influence the investigation
* Sun-tanned skin (important for the subgroup of subjects planned for Raman measurements)
* Regular use of tanning beds
* Any topical medication at the test area within the last 7 days prior to the start of the study
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. antiallergics) and/or within the last 7 days prior to the start of the study
* Past cosmetic surgery procedure in the test area (e.g. laser, facelift)
* Cosmetic surgery procedure in the test area, e.g. IPL (Intensed Pulsed Light), botox, chemical peel, dermabrasion within the last 2 years prior to the start of the study and/or throughout the entire course of the study
* Medical treatment for wrinkle reduction (e.g. peeling with vitamin A or fruit acids) on the face within the last 2 weeks prior to the start of the study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Anti-wrinkle efficacy will be assessed in the periorbital regions wrinkles using DermaTOP. Parameters measured: Rz and Ra, representing mainly the rough structure (Rz) or the finer skin structure (Ra). | 8-weeks

SECONDARY OUTCOMES:
Change from baseline in skin firmness by Cutometer [mm] after 2, 4 and 8 weeks | 8-weeks
Change from baseline in skin elasticity by Cutometer after 2, 4 and 8 weeks | 8-weeks
Change from baseline in skin hydration (assessed on skin capacitance by Corneometer [a.u.]) after 2, 4 and 8 weeks | 8-weeks
Change from baseline in skin barrier function (assessed on transepidermal waterloss by Tewameter [g/(m²h)]) after 2, 4, 8-weeks | 8-weeks
Change from baseline in ceramides by Raman Spectroscopy [a.u.] on a subgroup of n=12 subjects per test product group after 2, 4 and 8 weeks | 8-weeks
Change in Image grading (Photodocumentation via USR-Clip) for skin radiance (3 trained graders will rank each pair of images in a blinded fashion) after 2, 4 and 8 weeks | 8-weeks
Change in wrinkle scores (Photodocumentation via USR-Clip) for anti-wrinkle efficacy (3 trained graders will rank each pair of images at the area of the crow feet's in a blinded manner) | 8-weeks
Subjective Evaluation of product traits assessed via questionnaire after 2, 4 and 8 weeks | 8-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Klaus-Peter Wilhelm, MD, Study Chair — proDERM GmbH
Locations (1):
- proderm GmbH, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No